CLINICAL TRIAL: NCT06699160
Title: Post Market Clinical Follow-up Study on the Refobacin Revision-3 Bone Cement and Its Instrumentation
Brief Title: Refobacin Revision-3 Bone Cement Post-Market Study
Status: Withdrawn | Type: Observational
Why Stopped: The study was discontinued upon availability of relevant data through bespoke reporting, which fulfilled the study's primary objectives
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2021-28C
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Revision Arthroplasty
Keywords: revision surgery; bone cement; Refobacin Revision
MeSH Terms: interventions — Second-Look Surgery; Reoperation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

INTERVENTIONS:
Device: Revision arthroplasty — Hip or knee revision surgery resulting from aseptic loosening of the prosthesis and/or infection of the prosthesis by gentamicin and/or clindamycin sensitive strains.
  Other Names: Revision; Revision surgery

SUMMARY:
The goal of this post-market study is to confirm the safety, performance and clinical benefits of the Refobacin Revision-3 Bone Cement when used in knee or hip revision surgeries. This will be done by collecting information on:

* removal of any metal components of the hip or knee implants used in combination with the cement
* frequency and incidence of adverse events
* overall pain and functional performance, subject quality of life, and radiographic parameters

DETAILED DESCRIPTION:
Multicenter, retrospective and prospective, non-controlled Post-Market Clinical Follow-Up (PMCF) study involving orthopedic surgeons skilled in knee or hip arthroplasty procedures.

Patients will be enrolled prospectively or retrospectively (minimum 3 years after their surgery, depending on the availability of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older and skeletally mature.
* Patient is capable of understanding the surgeon's explanations and following his/her instructions, able and willing to participate in the follow-up program.
* Patient gave consent to take part in the study by signing the Ethics Committee approved Informed Consent Form (ICF).
* Patient who underwent or will undergo a hip or knee revision surgery with a Zimmer Biomet implant and the Refobacin® Revision-3 Bone Cement.
* Patient meets at least one of the following indications, as stated in the Instructions for Use (IFU):

  * Patients requires a revision operation resulting from aseptic loosening of the prosthesis and/or infection of the prosthesis by gentamicin and/or clindamycin sensitive strains.
  * Patients undergoing a two-stage revision that requires the fabrication and fixation of short-term total or hemi joint StageOne™ spacers. The device is intended for use in conjunction with systemic antimicrobial therapy (standard approach to an infection).

Additional inclusion criteria for patients receiving a StageOne™ spacer, as stated in the IFU:

* Implantation period of a maximum of 180 days.
* The molded temporary prosthesis is only indicated for patients who will consistently use traditional mobility assist devices (e.g. crutches, walkers) throughout the implant period.

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient is known to be pregnant or breastfeeding.
* Patient has any condition that would, in the judgment of the Investigator, place the patient at undue risk or interfere with the study.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant).
* Patient has plans to relocate during the study follow-up period.
* As stated in the IFU, patient with known hypersensitivity to gentamicin and/or clindamycin and/or to other constituents of the bone cement.
* Additional exclusion criteria for patients receiving a StageOne™ spacer, as stated in the IFU:

  * The infected Total Hip/Knee Replacement (THR/TKR) devices cannot be removed.
  * A systemic or secondary remote infection is expected or confirmed.
  * Lack of adequate bone structure precludes adequate support of the prosthesis in the proximal femur or acetabular region, or
  * Lack of adequate competence (anatomical and functional) of peripheral ligamentous apparatus and extensor mechanism.
  * The patient is sensitive (allergic) to aminoglycosides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population target is all subjects undergoing knee or hip revision surgeries with Refobacin® Revision-3 and a Zimmer Biomet implant approved for revision cases and who meet all of the inclusion and none of the exclusion criteria. Patients requiring a Zimmer Biomet StageOne™ spacer during a two-stage revision will be enrolled for subgroup analysis too.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 3, 5 and 10 years post-operatively
  * removal of any metal components of the hip or knee implants used in combination with the cement
  * frequency and incidence of adverse events

SECONDARY OUTCOMES:
EuroQuol 5D (EQ-5D) Score | 1, 3, 5 and 10 years post-operatively (retrospective, if available, or prospective)
  Subject quality of life assessed through the completion of an EQ-5D questionnaire, when available
Harris Hip Score / Knee Society Score | 1, 3, 5 and 10 years post-operatively (retrospective, if available, or prospective)
  Pain and functional performance assessed through the completion of an Harris Hips Score (HHS) or Knee Society Score (KSS) questionnaires, when available, depending on whether the revision procedure was performed on hip or knee
Radiographic evaluation | 1, 3, 5 and 10 years post-operatively (retrospective, if available, or prospective)
  Radiographic evaluation, when available, include but is not limited to: radiolucency, cement mantle, osteolysis, atrophy, hypertrophy, migration/subsidence and heterotopic ossification.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Clin Op Dir, Study Director — Zimmer Biomet
Locations (1):
- Diakonessenhuis UMC Utrecht, Utrecht, Netherlands